CLINICAL TRIAL: NCT03409718
Title: Comprehensive Shoulder System Database Retrieval
Brief Title: Database Retrieval for the Comprehensive Shoulder
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: ORTHO.CR.EX003
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Osteoarthritis of the Shoulder; Avascular Necrosis; Rheumatoid Arthritis; Prior Failed Revision; Correction of Functional Deformity; Fracture of Proximal End of Humerus; Cuff Tear Arthropathy
Keywords: Total Shoulder Arthroplasty; Medical Device; Performance; Safety; Shoulder Prosthesis
MeSH Terms: conditions — Osteonecrosis; Arthritis, Rheumatoid; Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Biomet Comprehensive Shoulder System: Subjects in need of a total shoulder arthroplasty who met the inclusion/exclusion criteria and received the Comprehensive Shoulder System.
  Interventions: Device: Biomet Comprehensive Shoulder System

INTERVENTIONS:
Device: Biomet Comprehensive Shoulder System — Total shoulder system designed to provide intraoperative flexibility for surgeons with unmatched humeral stem options, and infinite humeral head offset possibilities while meeting the growing demand for ease of glenoid preparation through a streamlined, low-profile, cannulated instrument platform

SUMMARY:
This study is a retrieval of database information regarding survivorship of the Comprehensive Shoulder System family of products. The primary objective of the retrieval is to collect data that will contribute to the post market surveillance requirements for this product and will provide feedback to design engineers, support marketing efforts and publications, and answer potential questions form reimbursement agencies.

DETAILED DESCRIPTION:
The Comprehensive Shoulder System has been cleared by the FDA via premarket notifications. No experimental or investigational surgical techniques or devices will be used in this study. All devices and products will be used in accordance with their instructions for use and/or approved labeling. The aim of the Comprehensive Shoulder System is to improve shoulder function and reduce pain.

One site will be used for this database retrieval. The number of patients involved will depend upon the size of the Comprehensive database available at Acromion, LLC.

ELIGIBILITY:
Inclusion Criteria:

* Must have one of the following indications:
* Non-inflammatory degenerative joint disease including osteoarthritis and avascular necrosis.
* Rheumatoid arthritis
* Revision where other devices or treatments have failed.
* Correction of functional deformity.
* Fractures of the proximal humerus, where other methods of treatment are deemed inadequate.
* Difficult clinical management problems, including cuff arthropathy, where other methods of treatment may not be suitable or may be inadequate.
* Need to obtain pain relief and improve function
* Ability and willingness of the patient to follow instructions, including control of weight and activity level
* A good nutritional state of the patient
* The patient must have reached full skeletal maturity

Exclusion Criteria:

* Absolute contraindications include infection, sepsis, and osteomyelitis.
* Uncooperative patient or patient with neurologic disorders who is incapable or unwilling to follow directions.
* Osteoporosis.
* Metabolic disorders which may impair bone formation.
* Osteomalacia.
* Distant foci of infections which may spread to the implant site.
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in need of a total shoulder arthroplasty which receive one of the devices in the Comprehensive Shoulder family and who meet all of the inclusion and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2011-02-24 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Implant survivorship is assessed counting the number of implant revisions | 10 years
  Implant survivorship will be documented by assessing the number of implant revisions occurring throughout the course of the study.

SECONDARY OUTCOMES:
Constant Shoulder Score | 10 years
  The Constant-Murley Shoulder Score is a scoring method used by clinicians to assess function of the shoulder. The standard score is on a scale of 0 to 100, with 0 being no shoulder function and 100 being excellent function.
Clinical Safety | 10 years
  Clinical safety is assessed through documentation of complications occurring during the course of the study.
Clinical Safety - Device Related | 10 years
  Clinical safety is assessed through documentation of device-related events occurring during the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Erin D Osborn, Study Director — Zimmer Biomet
Locations (1):
- Acromion LLC, Towson, Maryland, United States